CLINICAL TRIAL: NCT01151449
Title: A Phase II Study of RO4929097 (IND 109291) in Advanced, Metastatic, or Recurrent Triple Negative Invasive Breast Carcinoma
Brief Title: Gamma-secretase/Notch Signalling Pathway Inhibitor RO4929097 in Treating Patients With Advanced, Metastatic, or Recurrent Triple Negative Invasive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03135; NCI-2012-03135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-076 (Other: University Health Network-Princess Margaret Hospital); 8561 (Other: CTEP); N01CM00032 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Male Breast Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (gamma-secretase/Notch signalling pathway inhibitor) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II clinical trial studies how well gamma-secretase/Notch signalling pathway inhibitor RO4929097 works in treating patients with advanced, metastatic, or recurrent triple negative invasive breast cancer. Gamma-secretase/Notch signalling pathway inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the antitumour activity of RO4929097 in recurrent and/or metastatic triple negative breast cancer through co-primary endpoints of overall response rate (ORR) using RECIST and 6-month progression-free survival rate (PFS).

SECONDARY OBJECTIVES:

I. To assess the antitumour activity of RO4929097 through secondary endpoints including: duration of radiologic response, progression-free and overall survival rates within the protocol defined follow-up period.

II. To assess the safety and tolerability of single agent RO4929097 in breast cancer.

III. To explore expression of Notch biomarkers in triple negative breast cancer and potential interaction with RO4929097 response and toxicity.

IV. To evaluate the downstream effects of RO4929097 in advanced triple negative breast cancer.

OUTLINE:

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast carcinoma that is recurrent or metastatic; patients must have "triple negative" breast cancer, defined as estrogen/progesterone receptor negative (< 10% positive on IHC for the respective receptor) and HER2/neu negative (0 or 1+ on IHC or FISH-negative)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Prior adjuvant, neoadjuvant and unlimited lines of chemotherapy for metastatic disease will be permitted; there must be at least a 4-week interval since the last chemotherapy or investigational treatment and a 2-week interval since radiotherapy or surgery
* Life expectancy of greater than 12 weeks
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 90 g/L
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100x 10^9/L
* Total bilirubin =< 1.25 x upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 1.5 x upper limit of normal (=< 5 X if liver metastases)
* Serum creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min for patients with creatinine levels above institutional (using Crockcroft-Gault Formula)
* All radiology studies must be performed within 28 days prior to start of therapy
* No serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, psychiatric illness, or any other medical conditions that might be aggravated by treatment or limit compliance
* No active malignancy at any other site
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patients must be able to swallow pills
* The effects of RO4929097 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Notch signal pathway inhibitors are known to be teratogenic, if women of childbearing potential do not abstain from sexual activity (documentation that they have been abstinent from sexual activity at least 4 weeks prior to study entry) they must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry; women of childbearing potential be can either be abstinent or use two forms of contraception for the duration of study participation, and be either abstinent or use two forms of contraception for at least 12 months post-treatment; men must use condoms when sexually active with women for the duration of study participation and at least 12 months post-treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study; at least 2 weeks must have elapsed since any surgery or radiotherapy
* Patients may not be receiving any other investigational agents
* Patients with known symptomatic brain metastases are excluded; patients with controlled brain metastases (no radiographic progression following radiation and/or surgical treatment and no neurological signs or symptoms) will be allowed but must NOT be currently taking corticosteroids (e.g. dexamethasone) to control neurologic symptoms of brain metastases; patients with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by CT or MRI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients with suspicion of active Hepatitis A, B or C infection and a resulting positive serological result, or have a history of liver disease, or other forms of hepatitis / cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* Patients known to be HIV-positive who are on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with baseline (within 7days prior to starting study treatment) QTc > 450 msec (male) or QTc > 470 msec (female);

  * History of risk factors for QT interval prolongation, including, but not limited to family or personal history of long QT syndrome, recurrent syncope without known etiology or sudden unexpected death
  * History of torsade de pointes or other significant cardiac arrhythmias or the need for concomitant meds with known potential to prolong QT interval or antiarrhythmics
* Patients who have not recovered to < CTCAE grade 2 toxicities related to prior therapy are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Castro NP, Fedorova-Abrams ND, Merchant AS, Rangel MC, Nagaoka T, Karasawa H, Klauzinska M, Hewitt SM, Biswas K, Sharan SK, Salomon DS. Cripto-1 as a novel therapeutic target for triple negative breast cancer. Oncotarget. 2015 May 20;6(14):11910-29. doi: 10.18632/oncotarget.4182. PMID 26059540

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 51 [41 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Using RECIST
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From start of treatment until disease progression or removal from treatment.
Measure: Number; unit: participants
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 6
participants | 1

2. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the diameters of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Computed using the Kaplan-Meier method.
Time Frame: Time from start of study treatment to the date of first progression or death from any cause, whichever occurs first, assessed at 6 months
Population: Inadequate data for PFS estimates as only 6 patients were accrued in the study.
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: as for outcome 2
Time Frame: Time from start of study treatment to the date of first progression or death from any cause, whichever occurs first, assessed at 3 months
Population: Inadequate data for PFS estimates as only 6 patients were accrued in the study.
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Radiologic Response
Description: The duration of radiologic response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Measure: Number; unit: months
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 1
months | 6.9

5. Secondary Outcome: Overall Survival
Description: Computed using the Kaplan-Meier method.
Time Frame: Within the protocol defined follow-up period.
Population: Inadequate data for OS estimates as only 6 patients were accrued in the study.
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor) (N=6)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
DEATH NOS (General disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Gamma-secretase/Notch Signalling Pathway Inhibitor) (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ALLERGIC REACTION (Immune system disorders) | 1
ANEMIA (Blood and lymphatic system disorders) | 3
ANXIETY (Psychiatric disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
BREAST PAIN (Reproductive system and breast disorders) | 1
CHEST PAIN - CARDIAC (Cardiac disorders) | 1
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3
CREATININE INCREASED (Investigations) | 1
DEPRESSION (Psychiatric disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
EDEMA TRUNK (General disorders) | 1
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1
FATIGUE (General disorders) | 4
FEVER (General disorders) | 1
FLASHING LIGHTS (Eye disorders) | 1
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
GGT INCREASED (Investigations) | 1
HEADACHE (Nervous system disorders) | 2
HOT FLASHES (Vascular disorders) | 1
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1
HYPERTENSION (Vascular disorders) | 2
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3
HYPONATREMIA (Metabolism and nutrition disorders) | 2
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
LYMPHEDEMA (Vascular disorders) | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 5
MALABSORPTION (Gastrointestinal disorders) | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
OTHER (Eye disorders) | 2
PAIN (General disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
SKIN INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1
VOMITING (Gastrointestinal disorders) | 2
WEIGHT GAIN (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less